CLINICAL TRIAL: NCT05684328
Title: Narrow Band Imaging Versus White Light for the Detection and Miss of Sessile Serrated Lesions：a Multicenter，Random，Back-to-back Trial
Brief Title: Narrow Band Imaging Versus White Light for the Detection and Miss of Sessile Serrated Lesion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Hospital of Hebei Medical University (Other); Yantaishan Hospital (Unknown); The Second Affiliated Hospital of Guangzhou University of Chinese Medicine (Unknown); 900 Hospital of Joint Logistics Support Force of PLA (Other); Heilongjiang provincial hospital (Unknown); Ankang Central Hospital (Other); Nongken Jiansanjiang People Hospital of Heilongjiang Province (Unknown); Huadong Hospital (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Qilu Hospital of Shandong University (Other); Shandong First Medical University (Other); Air Force Military Medical University, China (Other); Tengzhou Central People's Hospital (Other Government); Chongqing General Hospital (Other); Haikou People's Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, MD,Director, Head of Department of Gastroenterology and Digestive Endoscopy Center, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NVWSDR-202212
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Sessile Serrated Lesion
Keywords: Sessile Serrated Lesions Miss Rate; Sessile Serrated Lesions Detection Rate; Narrow Band Imaging; Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLI Then NBI Withdrawal Group (Experimental): After successful intubation of the cecum, carefully inspect the whole colorectal mucosa by white light imaging(WLI) during the first colonoscopy withdraw. Then reinsert to the cecum and withdraw with narrow band imaging(NBI). Stop watch will be utilized to remind endoscopists.
  Interventions: Procedure: WLI Then NBI Withdrawal
- NBI Then WLI Withdrawal Group (Active Comparator): After successful intubation of the cecum, carefully inspect the whole colorectal mucosa by narrow band imaging(NBI) during the first colonoscopy withdraw. Then reinsert to the cecum and withdraw with white light imaging(WLI). Stop watch will be utilized to remind endoscopists.
  Interventions: Procedure: NBI Then WLI Withdrawal

INTERVENTIONS:
Procedure: WLI Then NBI Withdrawal — Patients in WLI then NBI withdrawal group will first be carefully inspected by white light imaging(WLI), each polyp found should be removed. According to the ESGE guideline of colorectal polypectomy, the lesions which size between 4-9mm should by removed by cold snare. Cold biopsy forceps could be utilized considering the difficulty in resection of flat and diminutive polyps(size ≤ 3mm). Then change to narrow band imaging(NBI) for the second withdraw to detect the lesions which found in second time but not the first.
  Arms: WLI Then NBI Withdrawal Group
Procedure: NBI Then WLI Withdrawal — Patients in NBI then WLI withdrawal group will first be carefully inspected by narrow band imaging(NBI), each polyp found should be removed. According to the ESGE guideline of colorectal polypectomy, the lesions which size between 4-9mm should by removed by cold snare. Cold biopsy forceps could be utilized considering the difficulty in resection of flat and diminutive polyps(size ≤ 3mm). Then change to white light imaging(WLI) for the second withdraw to detect the lesions which found in second time but not the first.
  Arms: NBI Then WLI Withdrawal Group

SUMMARY:
Narrow band imaging(NBI) could improve the detection of colorectal lesions, previous investigations demonstrated its potential in detecting not only colorectal adenoma but non-adenomatous polyps, including sessile serrated lesions. But no randomized controlled trials with NBI versus white light imaging(WLI) have been conducted to give a definitive conclusion with statistically significant differences. Therefore, we performed a multicenter, prospective, back to back, randomized controlled trial to compare sessile serrated lesions detection and miss rate of withdraw by NBI and WLI in colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age are between 45-85
* Patients who have indications for screening
* Patients who have signed inform consent form.

Exclusion Criteria:

* Patients who have undergone colonic resection
* Patients with alarming signs and symptoms of colorectal cancer: hematochezia, melena, anemia, weight loss, abdominal mass, positive digital rectal examination
* Patients with highly suspected or confirmed colorectal cancers by radiographic and laboratory tests
* Patients with abnormal blood coagulation or taking antiplatelets or anticoagulants within 7 days before colonoscopy
* Patients with inflammatory bowel diseases
* Patients with hereditary colorectal cancer syndrome (including familial adenomatous polyposis).
* Patients with pregnancy, severe chronic cardiopulmonary and renal disease.
* Patients with therapeutic colonoscopy for existing lesions
* Patients with failed cecal intubation
* Patients with poor bowel preparation quality that necessitated a second bowel preparation
* Patients refusing to participate or to provide informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
sessile serrated lesions miss rate(SSLMR) | 60 minutes
  Sessile serrated lesions(SSLs) detected in the second-pass examination were defined as missed SSLs; the sessile serrated lesions miss rate(SSLMR) was defined as follows: number of SSLs detected in the second-pass examination/total number of SSLs detected in both two pass.

SECONDARY OUTCOMES:
sessile serrated lesions detection rate(SSLDR) | 60 minutes
  Sessile serrated lesions detection rate(SSLDR) is the number of patients with at least one sessile serrated lesion detected by narrow band imaging or white light imaging, divided by the total number of patients.
adenoma miss rate(AMR) | 60 minutes
  Adenomas detected in the second-pass examination were defined as missed adenomas; the adenoma miss rate(AMR) was defined as follows: number of adenomas detected in the second-pass examination/total number of adenomas detected in the two pass.
adenoma detection rate(ADR) | 60 minutes
  Adenoma detection rate(ADR) is the number of patients with at least one adenoma detected by narrow band imaging or white light imaging, divided by the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zhao S, Song Y, Wang S, Wang R, Feng Z, Gong A, Yang X, Pan P, Yao D, Zhang J, Zhu Y, Li T, Bi J, Ren X, Tang X, Li Q, Yu D, Zheng J, Song B, Wang P, Chen W, Shang G, Xu Y, Xu P, Lai Y, Xu H, Yang X, Sheng J, Tao Y, Li X, Zhu Y, Zhang X, Shen H, Ma Y, Wang F, Wu L, Wang X, Li Z, Bai Y. Reduced Adenoma Miss Rate With 9-Minute vs 6-Minute Withdrawal Times for Screening Colonoscopy: A Multicenter Randomized Tandem Trial. Am J Gastroenterol. 2023 May 1;118(5):802-811. doi: 10.14309/ajg.0000000000002055. Epub 2022 Oct 11. PMID 36219172
- [Background] Li J, Zhang D, Wei Y, Chen K, Wu R, Peng K, Hou X, Li L, Huang C, Wang Y, Xun L, Xu H, Wang J, Chen Z, Shen M, Liu F. Colorectal Sessile Serrated Lesion Detection Using Linked Color Imaging: A Multicenter, Parallel Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2023 Feb;21(2):328-336.e2. doi: 10.1016/j.cgh.2022.03.033. Epub 2022 Apr 4. PMID 35390509
- [Background] Rex DK, Clodfelter R, Rahmani F, Fatima H, James-Stevenson TN, Tang JC, Kim HN, McHenry L, Kahi CJ, Rogers NA, Helper DJ, Sagi SV, Kessler WR, Wo JM, Fischer M, Kwo PY. Narrow-band imaging versus white light for the detection of proximal colon serrated lesions: a randomized, controlled trial. Gastrointest Endosc. 2016 Jan;83(1):166-71. doi: 10.1016/j.gie.2015.03.1915. Epub 2015 May 5. PMID 25952085
- [Derived] Wei J, Zhang S, Fang Q, Sui X, Tang X, Shi L, Zhao Y, Hu H, Huang Z, Huang X, Zhang H, Wang S, Li X, Wang C, Guo Y, Xu B, Wu W, Su Y, Chen L, Wei R, Li P, Shi L, Tang B, Qiao X, Xu M, Zhang J, Ji R, Ji D, Gong A, Li B, Ren J, Jiang Z, Xu H, Li M, Wang W, Yu J, Feng Z, Zhang J, Yao D, Li Z, Zhao S, Bai Y. Impact of Narrow-Band Imaging on Sessile Serrated Lesion Miss Rate: A Multicenter Randomized Tandem Colonoscopy Trial. Clin Gastroenterol Hepatol. 2026 Feb 2:S1542-3565(26)00055-8. doi: 10.1016/j.cgh.2026.01.027. Online ahead of print. PMID 41638419